CLINICAL TRIAL: NCT05700474
Title: Enhancing Wellness Through Affirming Services and Education
Acronym: EASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00111885
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: HIV; Mental Health Disorder; Substance Use
Keywords: HIV; Mental Health; Substance Use; PrEP; Comorbidity
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): There is one arm of the study and this involves participating in holistic behavioral health treatment for people living with HIV and the LGBTQ+ community for a 6 month period. Specific services include individual and group therapy, case management, peer support, and behavioral health education and awareness
  Interventions: Behavioral: Comprehensive outpatient behavioral health care

INTERVENTIONS:
Behavioral: Comprehensive outpatient behavioral health care — Participation will include clinical assessment and outpatient behavioral health services, case management, individual and group counseling, peer support, case management, and education regarding behavioral health and medical care
  Other Names: EASE

SUMMARY:
The goal of this treatment study is to learn about the mental health, substance use and physical health outcomes associated with participating in the EASE holistic behavioral health and wellness program for individuals identifying as LGBTQ+ and/or living with HIV. The main questions it aims to answer are:

1. Do important health outcomes, including substance use, mental health and social support related outcomes of individuals living with HIV and/or identifying as LGBTQ who participated in the holistic behavioral health and wellness program change after study participation?
2. Does a tailored approach to meet the specific needs of different subpopulations including 1) older (40+) PLWH and/or LGBTQ individuals with or at risk for additional health comorbidities and 2) PLWH and/or LGBTQ young adults (18-40) improve health outcomes including improvement in health and health behaviors .

Participants will be asked to:

* participate in 6 months of behavioral health treatment tailored to their needs, which may include individual counseling, group counseling, case management, peer support, and related education.
* Complete surveys at the time of study entry and 6 months later to measure changes in health outcomes over time.

DETAILED DESCRIPTION:
Enhancing Wellness through Affirming Services and Education (EASE) is a comprehensive behavioral health program aimed at improving health outcomes for individuals living with HIV and individuals in the LGBT community in Charlotte NC. Over the course of the proposed five-year program, 200 clients will receive an array of services to address substance use and mental health as well as underlying conditions including trauma, minority stress, comorbidities, stigma, and life instability (i.e. unstable housing, lack of access to medical care, employment barriers, and isolation).

EASE is a collaboration led by the Center for Health Policy and Inequalities Research with county and community partners including Mecklenburg County Community Support Services, RAIN, and individual therapists. Service offered will include evidence-based individual and group therapy, case management, peer programming, psychoeducation, and comorbidity management education. Building on previously successful programming, EASE will serve two client populations with tailored programs to meet their distinct needs. One track will serve an older population (over 40) with current drug use and living with or at higher risk of HIV to address substance use along with mental health and medical co-morbidities. A focus on overall wellness addressing stress management, nutrition, and chronic illness management will dovetail with substance use and mental health treatment to engage clients in whole body/mind wellness. The second track will serve minority LGBTQ+ adults, primarily adults under 40 to meet their specific mental and physical health needs addressing substance use, mental health, intersectional stress, gender-affirming health care, life skills development and sexual health . The LGBTQ+ community, particularly minority communities, has experienced more isolation and worse outcomes during the COVID pandemic; this track aims to address the behavioral health of this population by supporting overall wellbeing. Programmatic outcomes will be assessed through two secure online surveys completed by participants at baseline and six months after baseline.

ELIGIBILITY:
Inclusion Criteria:

1. HIV diagnosis or self-identified LGBTQ+
2. Any alcohol or illicit substance use in the last 90 days
3. 18 or older
4. Residing in Mecklenburg County or surrounding areas.

Exclusion Criteria:

1) Inability to consent for services due to reduced mental or physical capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms measured by the PHQ-9 | Baseline to 6 month follow-up survey
  PHQ-9 is a nine item depression scale with scores ranging from 0 to 27. A higher score indicates greater depressive symptoms
Change in anxiety symptoms measured by the Hospital Anxiety and Depression Scale (HADS) (Anxiety subsection) | Baseline to 6 month follow-up survey
  HADS anxiety subscale is a seven item anxiety scale with scores ranging from 0 to 21. A higher score indicates greater anxiety
Change in alcohol use as measured by alcohol use frequency questions | Baseline to 6 month follow-up survey
  The participant survey will include questions regarding any use of alcohol use in last 30 days and days of use in the last 30 days
Change in illicit substance use as measured by illicit substance use frequency questions | Baseline to 6 month follow-up survey
  The participant survey will include questions regarding any use of illicit drugs and 30 day use of illicit drugs

SECONDARY OUTCOMES:
Change in HIV-related stigma as measured by the HIV stigma scale | Baseline to 6 month follow-up survey
  The negative self-image subscale of HIV stigma scale has 13 items with likert response scores ranging from 13 to 52; higher scores indicate greater negative self image

CONTACTS AND LOCATIONS:
Overall Officials: Susan Reif, PhD, MSW, Principal Investigator — Duke University
Locations (1):
- Susan Reif, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No